CLINICAL TRIAL: NCT06585826
Title: Investigation the Urinary Incontinence Awareness of Syrian Women With Temporary Protection Status in Turkey
Brief Title: Urinary Incontinence Awareness of Syrian Women
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, PT, PhD, Karabuk University
Other Study IDs: Urinary incontinence Awareness
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Syrian female: Sociodemographic characteristics of women will be evaluated.
- Turkish female: Sociodemographic characteristics of women will be evaluated.

SUMMARY:
This study aimed to investigate the UI knowledge, attitudes, and awareness of Syrian females under temporary protection status in Turkey and compare it with Turkish females. Establishing societal standards surrounding urinary incontinence beliefs and attitudes can alter societal approaches to urinary incontinence. Early diagnosis and treatment can reduce the financial burden when urinary incontinence ceases to be an issue that needs to be hidden. Additionally, as females become more aware of urinary incontinence, urinary incontinence symptoms, urinary incontinence prevention, and treatment approaches, the number of patients receiving help for incontinence will increase.

DETAILED DESCRIPTION:
This study explores the knowledge, attitudes, and awareness of urinary incontinence (UI) among Syrian women under temporary protection in Turkey, compared to Turkish women. Involving 327 participants (186 Turkish, 141 Syrian), the study assesses sociodemographic data, gynecological and incontinence-related questions, and the Urinary Incontinence Awareness and Attitude Scale (URINAS). The study underscores the impact of sociocultural and economic factors on gender-specific health disorders, especially among refugees, and emphasizes the need for culture-specific interventions to enhance UI awareness among immigrant women. The findings can offer valuable insights for developing health policies and awareness programs aimed at improving UI management and reducing the stigma associated with it.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years of age
* volunteer for participation
* be under temporary protection

Exclusion Criteria:

* illiteracy
* any neurological disease that would affect cooperation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study was conducted with Syrian females under temporary protection status and Turkish females living in Karabuk between January 2024-May 2024. The study data was sent to individuals via e-mail.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Personal information form | Baseline
  Personel demographic and social information will be recorded used a form.
Urinary incontinence awareness and attitude scale | Baseline
  The scale consists of five sub-parameters: factors that prevent it from being accepted as a health problem, coping with UI, health motivation, restriction, and fear of UI. The answers given to each statement on the scale are in 5-point Likert type. The scale did not have a total score. Scores from sub-parameters: for the factors that prevent it from being accepted as a health problem sub-parameter (8-40); for the health motivation sub-parameter (5-25); for the coping with urinary incontinence subscale (6-30); for the restriction sub-parameter (3-15); It is (4-20) for the fear of UI subscale. On the basis of the median score, the incontinence awareness and attitude scale were interpreted as poor, moderate, or good.

CONTACTS AND LOCATIONS:
Overall Officials: Metehan Yana, PhD, Study Chair — Karabuk University
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van den Muijsenbergh ME, Lagro-Janssen TA. Urinary incontinence in Moroccan and Turkish women: a qualitative study on impact and preferences for treatment. Br J Gen Pract. 2006 Dec;56(533):945-9. PMID 17132383
- [Result] Roa L, Kent S, Yaskina M, Schulz J, Poirier A. Knowledge of pelvic floor disorders amongst immigrant women in Canada. Int Urogynecol J. 2021 Nov;32(11):3077-3084. doi: 10.1007/s00192-020-04662-1. Epub 2021 Feb 23. PMID 33620531
- [Result] Balsara ZP, Wu I, Marsh DR, Ihsan AT, Nazir R, Owoso E, Robinson C, Darmstadt GL. Reproductive tract disorders among Afghan refugee women attending health clinics in Haripur, Pakistan. J Health Popul Nutr. 2010 Oct;28(5):501-8. doi: 10.3329/jhpn.v28i5.6159. PMID 20941902